CLINICAL TRIAL: NCT06325540
Title: Clinical Success of Indirect Pulp Capping Using Biodentine, Theracal PT and Therabase in Primary Molars: 1-Year Follow-Up
Brief Title: Clinical Success of Indirect Pulp Capping: 1-Year Follow-Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pulpcapping
Record Dates: First submitted 2024-03-06; First posted 2024-03-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2024-03

CONDITIONS: Dentin, Carious; Indirect Pulp Capping
Keywords: calcium silicate; deep dentine carries; indirect pulp capping
MeSH Terms: conditions — Dental Caries | interventions — tricalcium silicate

STUDY DESIGN:
Intervention Model Description: Indirect pulp capping will be applied to primary molar teeth with deep dentin caries in 3 groups with 3 different materials(biodentine, thermal pt, therabase).
Who Masked: Participant, Outcomes Assessor
Masking Description: patients and the researcher who evaluates the follow-up results of the patients will not know which material was used for indirect pulp coating.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- theracal pt (Experimental): Teeth treated with indirect pulp capping with theracal pt
  Interventions: Procedure: indirect pulp capping with theracal pt
- therabase (Experimental): Teeth treated with indirect pulp capping with therabase
  Interventions: Procedure: indirect pulp capping with therabase
- biodentine (Active Comparator): Teeth treated with indirect pulp capping with biodentine
  Interventions: Procedure: indirect pulp capping with biodentine

INTERVENTIONS:
Procedure: indirect pulp capping with theracal pt — indirect pulp capping using the theracal pt material
  Arms: theracal pt
Procedure: indirect pulp capping with therabase — indirect pulp capping using the therabase material
  Arms: therabase
Procedure: indirect pulp capping with biodentine — indirect pulp capping using the biodentine material
  Arms: biodentine

SUMMARY:
The goal of this clinical trial is to compare the clinical success of theracal pt, therabase, and biodentine indirect pulp capping on primary molars with deep dentin caries. Indirect pulp capping was used on the primary molars of the participants with deep dentin caries. It is aimed to compare the success of biodentine, which is considered the gold standard used in capping treatments, and the currently marketed Teracal PT and Therabase materials after 1, 6 months and 1 year, with biodentine and with each other, and find out which material is more successful.

DETAILED DESCRIPTION:
This study utilized a parallel group, randomized controlled design and enrolled patients who visited the Department of Pediatric Dentistry, Health Sciences University, İstanbul, Turkey, in the period of 2020-2022. The study protocol was approved by the Health Sciences University Hamidiye Clinical Research Ethics Committee (7/34).

All procedures were conducted in accordance with the ethical standards of the relevant national and institutional committees on human experimentation with the Helsinki Declaration of 1975, as revised in 2013. The parents or legal guardians provided written in formed consent.

The sample size was calculated using a G*Power program (G*power 3.1 version) for the distribution of the success rates in the Biodentine, Therabase and TheraCal PT groups regarding the follow-up periods, the following parameters were used: medium effect size f 0.34, error = 0.05, minimum 80% power. Based on these parameters, the total sample size was calculated as 28 participants for each group.

This study was conducted as a prospective clinical and radiographic evaluation. A total of 76 teeth (first and second primary molars) from 5- to 9-year-old healthy and cooperative children with nonclinical and radiographic evidence of infection symptoms and with indications for indirect pulp treatment were included in this study. The teeth were divided into three groups according to the pulp capping materials.

Inclusion and exclusion criteria:

Healthy patients aged 5-9 years were recruited from the pediatric dental clinic at Health Sciences University. Based on the clinical and radiographic examinations, the inclusion criteria were previously untreated first and second primary molars in cooperative children with good general health, which had deep dentin caries involving occluso-proximal surfaces but showed positive response to vitality tests (electrical pulp test and cold stimulation) (Endo Ice, Hygienic; Coltene/Whaledent AG, Altst€atten, Switzerland and Diagnostic Unit; SybronEndo, Orange, CA); were radiographically detected with caries penetration involving approximately 3/4 of the dentin thickness; were considered to have a potential to result in pulp exposure when the entire caries was cleared according to the complete excavation procedure in which the end point of carious tissue removal is the hard dentin; and showed a moderate response to chemical and thermal stimuli. Clinical success criteria were as follows: signs of irreversible pulpitis (such as spontaneous pain, prolonged pain response), presence of percussion or palpation, pathological mobility, infectious symptoms such as fistula or abscess, and discoloration in the clinical examination. Radiographic success criteria included presence of radiolucency in the furcation or periapical regions, thickening of the periodontal spaces, and internal or external root resorption.

Clinical practice:

Two pediatric dentists screened each patient for inclusion and exclusion criteria during a preoperative oral examination and participants that met the inclusion criteria were randomly divided into three groups: Biodentine group (n =25), TheraCal PT group (n=26), Therabase group (n =25).

Following the application of topical and local anaesthesia injection (2% lidocaine hydrochloride with epinephrine 1:80,000; Septodont, Saint-Maur-des-Fosses, France), rubber-dam isolation (Dental Dam, Coltène Whaledent, Langenau, Germany) were performed. The tooth was disinfected by scrubbing with 2% chlorhexidine. The carious peripheral dentin was removed using a high-speed dental diamond bur (Dentsply, Dentsply Maillefer, Baillaigues, Switzerland) and the infected and necrotic soft dentin layer in the center was carefully removed to prevent pulp exposure. Cavity excavation was stopped when the residual dentin over the pulp tissue showed increased resistance to manual instrumentation, and the demineralized dentin (affected dentin) was left at the floor of the cavity. After removal of carious, the cavities were washed with 2% chlorhexidine gluconate irrigation solution (Klorhex, Drogsan, Türkiye) and then were dried with an air-water spray and cotton pellets. Biodentine, TheraCal PT and Therabase materials were applied according to the manufacturer's instructions.

Biodentine group: The entire residual demineralized dentin tissue covered with approximately 1mm tricalcium silicate pulp-capping material, Biodentine (Septodont,Saint-Maur-des-Fossés,France) by avoiding the placement of the material on enamel or margins of the cavity. After application of Biodentin, 12-min setting time was allowed for setting, in accordance with the recommendations of the manufacturer.

Theracal PT group: The entire residual demineralized dentin tissue covered with maximum thickness of 1mm flowable form of resin-modified calcium silicate-containing material, (TheraCal PT,Bisco Inc.,Schaumburg,IL,USA) by avoiding the placement of the material on enamel or margins of the cavity. After appllication of TheraCal PT, the polymerization for 20s (Elipar Deep Cure; 3 M ESPE, St. Paul, MN, USA), in accordance with the recommendations of the manufacturer.

Therabase group: The entire residual demineralized dentin tissue covered with maximum thickness of 1mm flowable form of dual-cured, calcium and fluoride releasing, self-adhesive base/liner material Therabase (Therabase PT,Bisco Inc.,Schaumburg,IL,USA) by avoiding the placement of the material on enamel or margins of the cavity. After appllication of TheraCal PT, the polymerization for 20s (Elipar Deep Cure; 3 M ESPE, St. Paul, MN, USA) in accordance with the recommendations of the manufacturer.

Afterwards, in all three groups, glass ionomer cement consisting of powder and liquid (Ketac Molar Easy Mix 3M ESPE, Germany) was placed on each capping material. Following the etching and bonding process, permanent restoration was finished with composite resin (Filtek Z250 Universal Restorative System, 3M ESPE DentalProducts, USA).

Clinical and radiographic examination: The patients were called for follow-up at 1 months, 6 months and 1 year during the first year. At each follow-up visit, a clinical examination was performed to assess the presence of tenderness to percussion or palpation, spontaneous pain or prolonged pain response, discoloration, infectious symptoms such as fistula or abscess, and pathological mobility. Additionally, a radiographic examination was performed to assess the presence of lesions in the furcation or periapical regions, internal or external root resorption, and thickening of the periodontal spaces. The teeth detected with at least one of these findings were considered 'unsuccessful.'

Statistical analysis All statistical analyses were performed by using software (SPSS, IBM SPSS Statistics 2022). Normality and homegenity of the data were evaluated by using Kolmogorov-Smirnov and Levene's Homogeneity tests. Pearson chi-square and Kruskall-Wallis H tests were performed to analyze data at the 95% confidence level (P = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 5-9 years
* Previously untreated first and second primary molars with deep caries
* First and second primary molar teeth with positive pulpal response in vitality tests
* Primary molar teeth with radiographically detected caries involving approximately ¾ of the dentin thickness
* Primary molar teeth with the potential for pulp exposure according to the procedure in which the carious tissue is completely removed

Exclusion Criteria:

* Teeth showing signs of irreversible pulpitis (spontaneous pain, no prolonged pain response)
* Teeth with symptoms of pain on percussion or palpation
* Teeth with pathological mobility
* Teeth with infectious symptoms such as fistula or abscess
* Teeth showing discoloration on clinical examination
* Radiolucency observed in the periapical region or furcation on radiographic examination

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
successful completion of research | 1 year
  Completion of 1-year follow-up of patients. The patients were called for follow-up at 1 months, 6 months and 1 year during the first year. At each follow-up visit, a clinical examination was performed to assess the presence of tenderness to percussion or palpation, spontaneous pain or prolonged pain response, discoloration, infectious symptoms such as fistula or abscess, and pathological mobility. Additionally, a radiographic examination was performed to assess the presence of lesions in the furcation or periapical regions, internal or external root resorption, and thickening of the periodontal spaces. The teeth detected with none of these findings at any time considered successful.
unseccessful completion of research | 1 year
  The patients were called for follow-up at 1 months, 6 months and 1 year during the first year. At each follow-up visit, a clinical examination was performed to assess the presence of tenderness to percussion or palpation, spontaneous pain or prolonged pain response, discoloration, infectious symptoms such as fistula or abscess, and pathological mobility. Additionally, a radiographic examination was performed to assess the presence of lesions in the furcation or periapical regions, internal or external root resorption, and thickening of the periodontal spaces. The teeth detected with at least one of these findings were considered 'unsuccessful.'

CONTACTS AND LOCATIONS:
Overall Officials: şükriye türkoğlu kayacı, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Sağlık Bilimleri Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No